CLINICAL TRIAL: NCT05907096
Title: A Phase 2, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study to Assess the Safety, Efficacy, and Tolerability of ARGX-117 in Improving Allograft Function in Recipients of a Deceased Donor Renal Allograft at Risk for Delayed Graft Function
Brief Title: ARGX-117 in Deceased Donor Kidney Transplant Recipients at Risk for Delayed Graft Function
Acronym: VARVARA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARGX-117-2201; 2022-503091-89-00 (Other: CTIS number)
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARGX-117 (Experimental): Patients receiving ARGX-117 intravenous infusions
  Interventions: Biological: ARGX-117
- Placebo (Placebo Comparator): Patients receiving placebo intravenous infusions
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARGX-117 — Intravenous administration of ARGX-117
  Arms: ARGX-117
Other: Placebo — Intravenous administration of placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety, efficacy and tolerability of ARGX-117 in Deceased Donor Kidney Transplant Recipients at Risk for Delayed Graft Function.

The study consists of 2 parts: part A comprises the main study period, and part B comprises the long-term observational follow-up period. During part A, after the screening period, eligible participants will be randomized to receive either ARGX-117 or placebo, entering the treatment and evaluation period (duration of up to 52 weeks). After the treatment period, participants will enter a follow-up period of up to 12 weeks.

The total study duration varies from approximately 64 weeks up to 5 years post-transplant depending on whether a participant enrols in part B of the study.

ELIGIBILITY:
Inclusion Criteria:

* Is at least the local legal age of consent for clinical studies and at least aged 18 years and less than 70 years
* Agree to use contraceptive measures consistent with local regulations
* Are diagnosed with ESRD and have been stable on chronic dialysis for at least 3 months
* Are recipients of de novo or second-time, single kidney transplant from a deceased donor, either DCD (donation after cardiac/circulatory death) or DBD ( (donation after brain death)
* Are ABO compatible with donor allograft, except for type A2 donor to type B recipient kidneys
* Have a negative cross match
* Have received pretransplant vaccinations for: Neisseria meningitidis, Streptococcus pneumoniae, and Haemophilus influenzae, or are willing to receive the vaccinations approximately 3 to 4 months posttransplant

Exclusion Criteria:

* Any history of prothrombotic disorder or history of thrombosis or hypercoagulable state, excluding vascular access clotting
* Any known history of complement deficiency
* Evidence of peritonitis in participants on peritoneal dialysis
* Received any solid organ, bone marrow, or hematopoietic stem cell transplant, with the exception of prior first kidney transplant
* High risk within the study period for recurrence of underlying renal disease in the opinion of the investigator
* Clinically significant comorbidity, recent major surgery (within 3 months of screening), history of any treatment nonadherence, or intention to have surgery during the study other than kidney transplantation; or any other medical condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Clinically significant active bacterial, viral, or fungal infection
* History of malignancy unless considered cured by adequate treatment, with no evidence of recurrence for 5 years or more before first study drug administration. Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer; Carcinoma in situ of the cervix; Carcinoma in situ of the breast; Incidental histological finding of prostate cancer
* History of current alcohol, drug, or medication abuse as assessed by the investigator
* Pregnant or lactating state or intention to become pregnant during the study

The full list of criteria can be found in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2024-02-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
eGFR at 24 weeks posttransplant | Up to 24 weeks
  Estimated glomerular filtration rate

SECONDARY OUTCOMES:
Proportion of participants with Delayed Graft Function (DGF) | Up to 52 weeks
Proportion of participants with fDGF | Up to 52 weeks
  Functional Delayed Graft Function
Duration of dialysis treatment for DGF within the first 30 days posttransplant | up to 30 days
Proportion of participants who have ongoing dialysis requirement at study day 31 | Up to 31 days
CRR at 72 hours posttransplant and on study day 8 | up to 8 days
  Creatinine reduction ratio
iBox score at 52 weeks posttransplant | up to 52 weeks
Dialysis-free participant survival through 52 weeks posttransplant | up to 52 weeks
(Death-censored) allograft survival through 52 weeks posttransplant | Up to 52 weeks
eGFR at 52 weeks posttransplant | up to 52 weeks
  Estimated glomerular filtration rate
Incidence of PNF | up to 12 weeks
  Primary Nonfunction
Serum concentrations for ARGX 117 | up to 64 weeks
Changes from baseline in free C2, total C2, and CH50 | up to 64 weeks
Incidence of anti-drug antibodies (ADA) against ARGX-117 | up to 64 weeks

CONTACTS AND LOCATIONS:
Locations (45):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Tampa General Hospital, Tampa, Florida
  - University of Illinois (UI) Health - Outpatient Care Center, Chicago, Illinois
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Columbia University, New York, New York
  - The Ohio State University, Columbus, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Monash Health - Monash Medical Centre, Clayton
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - Tirol Kliniken - A.o. Landeskrankenhaus Innsbruck, Innsbruck
  - Allgemeines Krankenhaus der Stadt Wien (AKH Wien), Vienna
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Brazil (5):
  - Centro Hospitalar e Universitario de Coimbra, Coimbra
  - Hospital Geral de Fortaleza, Fortaleza
  - Santa Casa de Misericordia de Porto Alegre - Hospital Dom Vicente Scherer, Porto Alegre
  - Hospital de Base, São Jose Do Rio Preto
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo (HC-FMUSP), São Paulo
- Canada (4):
  - Hôpital Maisonneuve-Rosemont - Centre de recherche, Montreal
  - McGill University Health Centre - Royal Victoria Hospital, Montreal
  - Vancouver Coastal Health - Vancouver General Hospital Diamond Healthcare Centre, Vancouver
  - Providence Health Care - St. Pauls Hospital, Vancouver
- France (6):
  - CHU Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Assistance Publique Hopitaux de Paris (AP-HP) - Hopital Henri Mondor, Créteil
  - CHU Grenoble Alpes - Hopital Michallon, La Tronche
  - Assistance Publique Hopitaux de Paris (AP-HP) - Hopital Necker-Enfants Malades, Paris
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - CHRU de Tours - Hopital Bretonneau, Tours
- Italy (3):
  - Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedale Universita Padova, Padua
  - Azienda Ospedaliero Universitaria Citta della Salute e della Scienza di Torino - Presidio Molinette, Torino
- Portugal (3):
  - Centro Hospitalar de Lisboa Ocidental EPE - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar Universitario Lisboa Central EPE - Hospital Curry Cabral, Lisbon
  - Centro Hospitalar Universitario de Santo Antonio, Porto
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol (HUGTP), Badalona
  - Hospital del Mar, Barcelona
  - Fundacio Puigvert, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves - Hospital General, Granada
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitari Doctor Peset, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided